CLINICAL TRIAL: NCT00792519
Title: Alcohol & HIV in Kenya: Stage 1 Trial of a Peer-Led Alcohol Behavior Intervention
Brief Title: Cognitive Behavioral Treatment to Reduce Alcohol Use Among HIV-Infected Kenyans
Acronym: KHBS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Moi Univeristy (Other); Indiana University School of Medicine (Other)
Responsible Party: Rebecca K Papas, PhD, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0703002442; R21AA016884 (NIH)
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-01

CONDITIONS: Binge Drinking; Alcohol Abuse; Alcohol Dependence; HIV Infections
Keywords: alcohol use; HIV; cognitive behavioral treatment; Kenya; hazardous/binge drinking; alcohol abuse/dependence
MeSH Terms: conditions — Binge Drinking; Alcoholism; HIV Infections; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT (Experimental): group cognitive behavioral treatment
  Interventions: Behavioral: CBT
- HIV support group (Active Comparator): group support
  Interventions: Behavioral: HIV support group

INTERVENTIONS:
Behavioral: HIV support group — group support
  Arms: HIV support group
Behavioral: CBT — group cognitive behavioral treatment
  Arms: CBT

SUMMARY:
This study will determine whether a cognitive behavioral intervention that demonstrates strong evidence in the U.S. of reducing alcohol use is effective when delivered by paraprofessionals in Kenya and compared against a usual care support group.

DETAILED DESCRIPTION:
Alcohol use and abuse have been associated with increased risky sexual behavior, poor adherence to antiretroviral therapy (ARVs) and toxicity from ARVs among those with HIV infection. As such, alcohol use and abuse have a major impact on HIV transmission and disease progression. Because alcohol abuse is widespread in Kenya, with estimates of hazardous drinking as high as 68% in general medicine clinics and 53% in HIV clinics, this Stage 1 pilot project will develop and evaluate a paraprofessionally led group cognitive behavioral treatment (CBT) targeting alcohol use among HIV infected Kenyans who were initiated on ARV therapy in the past year. Although CBT is well-suited to the Kenyan setting because it is comparatively structured and consistent with the Kenyan conceptual model of drinking behavior, it requires adaptation for group paraprofessional delivery due to the extremely limited supply of Kenyan mental health professionals. The goal of this 24-month capacity-building R21 study is to evaluate the efficacy of a novel application of CBT, a 6-session paraprofessionally led group in Eldoret, Kenya, when compared against a usual care support group, to reduce hazardous and binge drinking among adult persons infected with HIV. This work will be conducted via the Kenya-U.S. HIV and Alcohol Research and Prevention Partnership-an experienced team of Kenyan and U.S. physicians, behavioral scientists, recovered substance users and persons infected with HIV. The team expands on well-established ties between the Academic Model for Providing Access to Health Care (AMPATH) and the Veterans Aging Cohort Study (VACS), a longitudinal clinical study of HIV and alcohol. AMPATH treats more than 65,000 HIV patients in 19 clinics in western Kenya. Our goals are to: 1) train Kenyan staff and investigators in research methods and train paraprofessionals in group CBT delivery; 2) pilot the CBT adaptation; and 3) evaluate the feasibility of the paraprofessionally led group CBT via a Stage 1 trial in which 56 HIV infected Kenyans are randomized to same-sex CBT or usual care HIV support groups.

ELIGIBILITY:
Inclusion Criteria:

* HIV outpatient
* hazardous or binge drinker
* drank any alcohol in past month
* ARV-eligible or initiated on ARVs in past 12 months
* within 1 hour travel distance of Eldoret, Kenya HIV clinic
* speak Kiswahili

Exclusion Criteria:

* active psychosis or suicidality
* plans to move within next 6 months > 1 hr travel distance from Eldoret HIV clinic
* physically unable to attend sessions
* ever attended AMPATH alcohol support group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
quantity and frequency of alcohol use | 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca K Papas, PhD, Principal Investigator — Brown University
Locations (1):
- AMPATH Centre, Eldoret, Rift Valley, Kenya

REFERENCES:
- [Background] Papas RK, Sidle JE, Martino S, Baliddawa JB, Songole R, Omolo OE, Gakinya BN, Mwaniki MM, Adina JO, Nafula T, Owino-Ong'or WD, Bryant KJ, Carroll KM, Goulet JL, Justice AC, Maisto SA. Systematic cultural adaptation of cognitive-behavioral therapy to reduce alcohol use among HIV-infected outpatients in western Kenya. AIDS Behav. 2010 Jun;14(3):669-78. doi: 10.1007/s10461-009-9647-6. PMID 19967441
- [Background] Papas RK, Sidle JE, Wamalwa ES, Okumu TO, Bryant KL, Goulet JL, Maisto SA, Braithwaite RS, Justice AC. Estimating alcohol content of traditional brew in Western Kenya using culturally relevant methods: the case for cost over volume. AIDS Behav. 2010 Aug;14(4):836-44. doi: 10.1007/s10461-008-9492-z. Epub 2008 Nov 18. PMID 19015972
- [Result] Papas RK, Sidle JE, Gakinya BN, Baliddawa JB, Martino S, Mwaniki MM, Songole R, Omolo OE, Kamanda AM, Ayuku DO, Ojwang C, Owino-Ong'or WD, Harrington M, Bryant KJ, Carroll KM, Justice AC, Hogan JW, Maisto SA. Treatment outcomes of a stage 1 cognitive-behavioral trial to reduce alcohol use among human immunodeficiency virus-infected out-patients in western Kenya. Addiction. 2011 Dec;106(12):2156-66. doi: 10.1111/j.1360-0443.2011.03518.x. Epub 2011 Aug 18. PMID 21631622
- [Derived] Galarraga O, Gao B, Gakinya BN, Klein DA, Wamai RG, Sidle JE, Papas RK. Task-shifting alcohol interventions for HIV+ persons in Kenya: a cost-benefit analysis. BMC Health Serv Res. 2017 Mar 28;17(1):239. doi: 10.1186/s12913-017-2169-4. PMID 28351364